CLINICAL TRIAL: NCT03262103
Title: Phase I Study of In Situ Autologous Vaccination Against Prostate Cancer With Intratumoral and Systemic Hiltonol® (Poly-ICLC) Prior To Radical Prostatectomy
Brief Title: Neoadjuvant Hiltonol® (PolyICLC) for Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ashutosh Kumar Tewari (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ashutosh Kumar Tewari, Professor, System Chairman of the Department of Urology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-2081
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Gleason 7-10; Immunotherapy; Neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — poly ICLC; Injections, Intramuscular

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Intratumoral (IT) Poly ICLC 0.5 mg IT once/week (week 1) Intramuscular (IM) Poly ICLC 1 mg IM twice weekly (weeks 3-6) Followed by Radical Prostatectomy at Week 10
  Interventions: Biological: Intratumoral (IT) Poly ICLC 0.5 mg; Biological: Intramuscular (IM) Poly ICLC; Procedure: Radical Prostatectomy
- Cohort 2 (Experimental): Intratumoral (IT) Poly ICLC 0.5 mg IT once/week (week 1+2) Intramuscular (IM) Poly ICLC 1 mg IM twice weekly (weeks 3-6) Followed by Radical Prostatectomy at Week 10
  Interventions: Biological: Intratumoral (IT) Poly ICLC 0.5 mg; Biological: Intramuscular (IM) Poly ICLC; Procedure: Radical Prostatectomy
- Cohort 3 (Experimental): Intratumoral (IT) Poly ICLC 1.0 mg IT once/week (week 1) Intramuscular (IM) Poly ICLC 1 mg IM twice weekly (weeks 3-6) Followed by Radical Prostatectomy at Week 10
  Interventions: Biological: Intratumoral (IT) Poly ICLC 1.0 mg; Biological: Intramuscular (IM) Poly ICLC; Procedure: Radical Prostatectomy
- Cohort 4 (Experimental): Intratumoral (IT) Poly ICLC 1.0 mg IT once/week (week 1+2) Intramuscular (IM) Poly ICLC 1 mg IM twice weekly (weeks 3-6) Followed by Radical Prostatectomy at Week 10
  Interventions: Biological: Intratumoral (IT) Poly ICLC 1.0 mg; Biological: Intramuscular (IM) Poly ICLC; Procedure: Radical Prostatectomy

INTERVENTIONS:
Biological: Intratumoral (IT) Poly ICLC 0.5 mg — 0.5 mg IT once/week (week 1)
  Arms: Cohort 1; Cohort 2
Biological: Intratumoral (IT) Poly ICLC 1.0 mg — 1.0 mg IT once/week (week 1)
  Other Names: Polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose
  Arms: Cohort 3; Cohort 4
Biological: Intramuscular (IM) Poly ICLC — 1 mg IM twice weekly (weeks 3-6)
  Other Names: Polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose
Procedure: Radical Prostatectomy — as per standard care

SUMMARY:
The purpose of this study is to test an approach of stimulating the body's immune system to attack prostate cancer. This study will test injection of a substance polylysine and carboxymethylcellulose (Poly-ICLC, Hiltonol®)through a needle guided by MRI (magnetic resonance imaging) ultrasound fusion technology into the prostate gland. Poly ICLC has been used to help the body in its fight against cancer. The first aim of the study is to determine the highest dose of a substance Poly-ICLC (Hiltonol®) that can be safely tolerated by the study participants. The second aim of the study is to find out the toxicity or side effects of poly-ICLC.

DETAILED DESCRIPTION:
This is a pilot dose escalation study of IT/IM Poly-ICLC in patients with high risk clinically localized prostate cancer. The dose and frequency of IT injections will be increased in successive cohorts to define a safe dose and schedule for further testing.

Intratumoral + intramuscular poly-ICLC in patients with clinical localized prostate cancer. In the current pilot clinical trial, poly-ICLC will be administered intratumorally (Artemis guided) and intramuscularly (e.g., deltoid muscle) prior to prostatectomy in patients with clinically localized prostate cancer. Based on the available preclinical data exploring intratumoral administration of PAMPs described above, we expect this approach will result in three immunomodulatory steps26:

Immunomodulatory Step 1: Innate immune local tumor killing induced by intratumoral poly-ICLC - the initial intratumoral injections are expected to induce activation/recruitment of IL-12, TNF-α, and other cytokines and NK cells, resulting in early tumor killing and antigen release.9-11 Poly-ICLC may also have a direct antiproliferative effect on tumor cells mediated by interferon-inducible nuclear enzyme systems.

Immunomodulatory Step 2: Th1 and cytotoxic T lymphocyte priming as a result of the repeated in-situ poly-ICLC 'danger signal' combined with the tumor antigens released in step 1 and further processed and cross-presented by poly-ICLC-activated myeloid dendritic cells.7,8 Poly-ICLC is expected to recruit myeloid dendritic cells and macrophages to the tumor site where they can load with antigens being released through the innate mechanisms, present them Th1 cells, and cross-present them to CD8 T cells in the tumor or in the regional lymph nodes, thus generating antigen specific cytotoxic T lymphocytes.

Immunomodulatory Step 3 (or "Boost" phase): Maintenance of the systemic anti-tumor immune response and migration of cytotoxic T lymphocytes to remote metastases, through repeated intramuscular poly-ICLC induction of chemokines, other costimulatory factors, and inflammasome activation.23-25 The rationale for followup with intramuscular maintenance is that as part of the comprehensive response, dsRNAs such as poly-ICLC induce various chemokines and costimulatory factors that help target the response to tumor. For example, one of these costimulatory factors is OX40, which belongs to the tumor necrosis factor family of cytokines, and helps maintain cytotoxic lymphocyte longevity and action at the tumor and metastatic sites.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 14 days prior to being registered for protocol therapy (Study Procedure Manual).
* Histologically confirmed adenocarcinoma of the prostate (with previous diagnostic tissue available for tumor marker analysis).
* Gleason 7 - 10, cT2a - cT3b adenocarcinoma of the prostate with plans for radical prostatectomy
* PSA ≥ 4 ng/ml
* Tumor visible on multiparametric MRI
* Tolerated previous transrectal ultrasound guided biopsy procedure under local anesthetic
* Uncomplicated previous TRUS biopsy procedure (i.e., no prior hospitalization due to sepsis, prostatic abscess or severe hemorrhage following TRUS prostate biopsy)
* Willing to undergo the intra-tumoral (IT) injection of the Poly-ICLC into the prostatic tumor as per the protocol
* No prior hormonal therapy with the exception of oral 5-alpha-reductase inhibitors (finasteride, dutasteride, etc.). Patients who have received prior oral anti-androgen therapies (bicalutamide, flutamide, nilutamide, etc.) must be off treatment for at least 6 weeks prior to enrollment. Patients who have received prior LHRH agonist or antagonist therapy (leuprolide, goserelin acetate, etc.) are eligible provided serum testosterone is > 50 mg/dl.
* No prior radiation therapy (external beam or brachytherapy) to the pelvis or prostate.
* No clinically significant infections as judged by the treating investigator.
* No characteristics suggesting a potential higher risk of infection with intraprostatic injections:

  * Recurrent urinary tract infections or history of prostatitis within 3 months prior to enrollment into the study.
  * Urine analysis positive for nitrites and leucocyte esterase. Such patients could be considered for the study after treatment and resolution of the infection.
  * Active proctitis
  * History of prostatic abscess
  * Taking immunosuppressive medication including systemic corticosteroids
  * Active hematologic malignancy
* No uncontrolled angina, congestive heart failure or MI within 6 months.
* Patients with history of HIV (if CD4+ T cell counts are ≥350 cells/µL on established ART therapy), Hepatitis B (with viral load below limits of quantification) or Hepatitis C (who have completed a curative therapy and have a viral load below the limit of quantification) are eligible for this study.
* No treatment with any investigational agent for any medical condition within 28 days prior to being registered for protocol therapy.

  * Adequate end organ function as determined by the following laboratory values:

    * White blood cell count (WBC) > 2.5 k/mm3
    * Absolute neutrophil count (ANC) > 1.5 k/mm3
    * Hemoglobin (Hgb) > 8.0 g/dL
    * Platelets > 100 k/mm3
    * Calculated creatinine clearance of > 60 cc/min using the Cockcroft-Gault formula:

Males: (140 - Age in years) × Actual Body Weight in kg 72 × Serum Creatinine (mg/dL)

* Bilirubin < 2.0 x ULN
* Aspartate aminotransferase (AST) < 2.5 x ULN
* Alanine aminotransferase (ALT) < 2.5 x ULN 18) Able to speak, read and write in English.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity level | Week 6
  3+3 dose escalation rules to define a safe dose of preoperative intratumoral (IT) plus intramuscular (IM) Polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose (poly-ICLC, Hiltonol®) prior to radical prostatectomy

SECONDARY OUTCOMES:
Number of adverse events | Week 6
  Safety as determined by the frequency of adverse events as per the Common Terminology for Adverse Events (CTCAE) version 4.0.
Time to PSA progression | up to Week 12
  The time to prostate-specific antigen (PSA) progression will be defined as the time to PSA > 0.2 ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh K. Tewari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sujit S Nair, Ph.D., Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Pound CR, Partin AW, Eisenberger MA, Chan DW, Pearson JD, Walsh PC. Natural history of progression after PSA elevation following radical prostatectomy. JAMA. 1999 May 5;281(17):1591-7. doi: 10.1001/jama.281.17.1591. PMID 10235151
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Sonpavde G, Di Lorenzo G, Higano CS, Kantoff PW, Madan R, Shore ND. The role of sipuleucel-T in therapy for castration-resistant prostate cancer: a critical analysis of the literature. Eur Urol. 2012 Apr;61(4):639-47. doi: 10.1016/j.eururo.2011.10.027. Epub 2011 Oct 24. PMID 22036643
- [Background] Levy HB, Levine AS. Antitumor effects of interferon and poly ICLC, and their possible utility as anti-neoplastic agents in man. Tex Rep Biol Med. 1981-1982;41:653-62. No abstract available. PMID 6189230
- [Background] Caskey M, Lefebvre F, Filali-Mouhim A, Cameron MJ, Goulet JP, Haddad EK, Breton G, Trumpfheller C, Pollak S, Shimeliovich I, Duque-Alarcon A, Pan L, Nelkenbaum A, Salazar AM, Schlesinger SJ, Steinman RM, Sekaly RP. Synthetic double-stranded RNA induces innate immune responses similar to a live viral vaccine in humans. J Exp Med. 2011 Nov 21;208(12):2357-66. doi: 10.1084/jem.20111171. Epub 2011 Nov 7. PMID 22065672
- [Background] Zhu X, Fallert-Junecko BA, Fujita M, Ueda R, Kohanbash G, Kastenhuber ER, McDonald HA, Liu Y, Kalinski P, Reinhart TA, Salazar AM, Okada H. Poly-ICLC promotes the infiltration of effector T cells into intracranial gliomas via induction of CXCL10 in IFN-alpha and IFN-gamma dependent manners. Cancer Immunol Immunother. 2010 Sep;59(9):1401-9. doi: 10.1007/s00262-010-0876-3. Epub 2010 Jun 12. PMID 20549206
- [Background] Okada H, Kalinski P, Ueda R, Hoji A, Kohanbash G, Donegan TE, Mintz AH, Engh JA, Bartlett DL, Brown CK, Zeh H, Holtzman MP, Reinhart TA, Whiteside TL, Butterfield LH, Hamilton RL, Potter DM, Pollack IF, Salazar AM, Lieberman FS. Induction of CD8+ T-cell responses against novel glioma-associated antigen peptides and clinical activity by vaccinations with alpha-type 1 polarized dendritic cells and polyinosinic-polycytidylic acid stabilized by lysine and carboxymethylcellulose in patients with recurrent malignant glioma. J Clin Oncol. 2011 Jan 20;29(3):330-6. doi: 10.1200/JCO.2010.30.7744. Epub 2010 Dec 13. PMID 21149657
- [Background] Chew V, Tow C, Huang C, Bard-Chapeau E, Copeland NG, Jenkins NA, Weber A, Lim KH, Toh HC, Heikenwalder M, Ng IO, Nardin A, Abastado JP. Toll-like receptor 3 expressing tumor parenchyma and infiltrating natural killer cells in hepatocellular carcinoma patients. J Natl Cancer Inst. 2012 Dec 5;104(23):1796-807. doi: 10.1093/jnci/djs436. Epub 2012 Nov 29. PMID 23197495
- [Background] Sivori S, Falco M, Della Chiesa M, Carlomagno S, Vitale M, Moretta L, Moretta A. CpG and double-stranded RNA trigger human NK cells by Toll-like receptors: induction of cytokine release and cytotoxicity against tumors and dendritic cells. Proc Natl Acad Sci U S A. 2004 Jul 6;101(27):10116-21. doi: 10.1073/pnas.0403744101. Epub 2004 Jun 24. PMID 15218108
- [Background] North RJ, Dunn PL, Havell EA. A role for tumor necrosis factor in poly(I:C)-induced hemorrhagic necrosis and T-cell-dependent regression of a murine sarcoma. J Interferon Res. 1991 Dec;11(6):333-40. doi: 10.1089/jir.1991.11.333. PMID 1839310
- [Background] Bogunovic D, Manches O, Godefroy E, Yewdall A, Gallois A, Salazar AM, Marie I, Levy DE, Bhardwaj N. TLR4 engagement during TLR3-induced proinflammatory signaling in dendritic cells promotes IL-10-mediated suppression of antitumor immunity. Cancer Res. 2011 Aug 15;71(16):5467-76. doi: 10.1158/0008-5472.CAN-10-3988. Epub 2011 Jul 5. PMID 21730023
- [Background] Black PL, Hartmann D, Pennington R, Phillips H, Schneider M, Tribble HR, Talmadge JE. Effect of tumor burden and route of administration on the immunotherapeutic properties of polyinosinic-polycytidylic acid stabilized with poly-L-lysine in carboxymethyl cellulose [Poly(I,C)-LC]. Int J Immunopharmacol. 1992 Nov;14(8):1341-53. doi: 10.1016/0192-0561(92)90005-6. PMID 1464467
- [Background] Kajiwara K, Morishima H, Akiyama K, Yanagihara Y. Expression and function of the inducible costimulator ligand B7-H2 in human airway smooth muscle cells. Allergol Int. 2009 Dec;58(4):573-83. doi: 10.2332/allergolint.09-OA-0113. Epub 2009 Sep 25. PMID 19776675
- [Background] Stevenson HC, Abrams PG, Schoenberger CS, Smalley RB, Herberman RB, Foon KA. A phase I evaluation of poly(I,C)-LC in cancer patients. J Biol Response Mod. 1985 Dec;4(6):650-5. PMID 2418163
- [Background] Hawkins MJ, Levin M, Borden EC. An Eastern Cooperative Oncology Group phase I-II pilot study of polyriboinosinic-polyribocytidylic acid poly-L-lysine complex in patients with metastatic malignant melanoma. J Biol Response Mod. 1985 Dec;4(6):664-8. PMID 2418164
- [Background] Krown SE, Kerr D, Stewart WE 2nd, Field AK, Oettgen HF. Phase I trials of poly(I,C) complexes in advanced cancer. J Biol Response Mod. 1985 Dec;4(6):640-9. PMID 2418162
- [Background] Hartman LL, Crawford JR, Makale MT, Milburn M, Joshi S, Salazar AM, Hasenauer B, VandenBerg SR, MacDonald TJ, Durden DL. Pediatric phase II trials of poly-ICLC in the management of newly diagnosed and recurrent brain tumors. J Pediatr Hematol Oncol. 2014 Aug;36(6):451-7. doi: 10.1097/MPH.0000000000000047. PMID 24309609
- [Background] Sabbatini P, Tsuji T, Ferran L, Ritter E, Sedrak C, Tuballes K, Jungbluth AA, Ritter G, Aghajanian C, Bell-McGuinn K, Hensley ML, Konner J, Tew W, Spriggs DR, Hoffman EW, Venhaus R, Pan L, Salazar AM, Diefenbach CM, Old LJ, Gnjatic S. Phase I trial of overlapping long peptides from a tumor self-antigen and poly-ICLC shows rapid induction of integrated immune response in ovarian cancer patients. Clin Cancer Res. 2012 Dec 1;18(23):6497-508. doi: 10.1158/1078-0432.CCR-12-2189. Epub 2012 Oct 2. PMID 23032745
- [Background] Rosenfeld MR, Chamberlain MC, Grossman SA, Peereboom DM, Lesser GJ, Batchelor TT, Desideri S, Salazar AM, Ye X. A multi-institution phase II study of poly-ICLC and radiotherapy with concurrent and adjuvant temozolomide in adults with newly diagnosed glioblastoma. Neuro Oncol. 2010 Oct;12(10):1071-7. doi: 10.1093/neuonc/noq071. Epub 2010 Jul 8. PMID 20615924
- [Background] Morse MA, Chapman R, Powderly J, Blackwell K, Keler T, Green J, Riggs R, He LZ, Ramakrishna V, Vitale L, Zhao B, Butler SA, Hobeika A, Osada T, Davis T, Clay T, Lyerly HK. Phase I study utilizing a novel antigen-presenting cell-targeted vaccine with Toll-like receptor stimulation to induce immunity to self-antigens in cancer patients. Clin Cancer Res. 2011 Jul 15;17(14):4844-53. doi: 10.1158/1078-0432.CCR-11-0891. Epub 2011 Jun 1. PMID 21632857
- [Background] Mangsbo SM, Ninalga C, Essand M, Loskog A, Totterman TH. CpG therapy is superior to BCG in an orthotopic bladder cancer model and generates CD4+ T-cell immunity. J Immunother. 2008 Jan;31(1):34-42. doi: 10.1097/CJI.0b013e3181587d29. PMID 18157010
- [Background] Houot R, Levy R. T-cell modulation combined with intratumoral CpG cures lymphoma in a mouse model without the need for chemotherapy. Blood. 2009 Apr 9;113(15):3546-52. doi: 10.1182/blood-2008-07-170274. Epub 2008 Oct 21. PMID 18941113
- [Background] Davies ME, Field AK. Effect of poly I:C/poly-L-lysine (poly ICL) on the development of murine osteogenic sarcoma. J Interferon Res. 1983;3(1):89-95. doi: 10.1089/jir.1983.3.89. PMID 6573430
- [Background] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067
- [Background] Salazar AM, Erlich RB, Mark A, Bhardwaj N, Herberman RB. Therapeutic in situ autovaccination against solid cancers with intratumoral poly-ICLC: case report, hypothesis, and clinical trial. Cancer Immunol Res. 2014 Aug;2(8):720-4. doi: 10.1158/2326-6066.CIR-14-0024. Epub 2014 May 6. PMID 24801836
- [Background] Maluish AE, Reid JW, Crisp EA, Overton WR, Levy H, Foon KA, Herberman RB. Immunomodulatory effects of poly(I,C)-LC in cancer patients. J Biol Response Mod. 1985 Dec;4(6):656-63. PMID 4087034
- [Background] Pilaro AM, Taub DD, McCormick KL, Williams HM, Sayers TJ, Fogler WE, Wiltrout RH. TNF-alpha is a principal cytokine involved in the recruitment of NK cells to liver parenchyma. J Immunol. 1994 Jul 1;153(1):333-42. PMID 8207246
- [Background] Morgan ET, Norman CA. Pretranslational suppression of cytochrome P-450h (IIC11) gene expression in rat liver after administration of interferon inducers. Drug Metab Dispos. 1990 Sep-Oct;18(5):649-53. PMID 1706245
- [Background] Salazar AM, Levy HB, Ondra S, Kende M, Scherokman B, Brown D, Mena H, Martin N, Schwab K, Donovan D, Dougherty D, Pulliam M, Ippolito M, Graves M, Brown H, Ommaya A. Long-term treatment of malignant gliomas with intramuscularly administered polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose: an open pilot study. Neurosurgery. 1996 Jun;38(6):1096-103; discussion 1103-4. PMID 8727138
- [Background] Butowski N, Chang SM, Junck L, DeAngelis LM, Abrey L, Fink K, Cloughesy T, Lamborn KR, Salazar AM, Prados MD. A phase II clinical trial of poly-ICLC with radiation for adult patients with newly diagnosed supratentorial glioblastoma: a North American Brain Tumor Consortium (NABTC01-05). J Neurooncol. 2009 Jan;91(2):175-82. doi: 10.1007/s11060-008-9693-3. Epub 2008 Sep 17. PMID 18797818
- [Background] Butowski N, Lamborn KR, Lee BL, Prados MD, Cloughesy T, DeAngelis LM, Abrey L, Fink K, Lieberman F, Mehta M, Ian Robins H, Junck L, Salazar AM, Chang SM. A North American brain tumor consortium phase II study of poly-ICLC for adult patients with recurrent anaplastic gliomas. J Neurooncol. 2009 Jan;91(2):183-9. doi: 10.1007/s11060-008-9705-3. Epub 2008 Oct 11. PMID 18850068
- [Background] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Background] Rothke M, Blondin D, Schlemmer HP, Franiel T. [PI-RADS classification: structured reporting for MRI of the prostate]. Rofo. 2013 Mar;185(3):253-61. doi: 10.1055/s-0032-1330270. Epub 2013 Feb 12. German. PMID 23404430
- [Background] Rosenkrantz AB, Lim RP, Haghighi M, Somberg MB, Babb JS, Taneja SS. Comparison of interreader reproducibility of the prostate imaging reporting and data system and likert scales for evaluation of multiparametric prostate MRI. AJR Am J Roentgenol. 2013 Oct;201(4):W612-8. doi: 10.2214/AJR.12.10173. PMID 24059400
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Gnjatic S, Ritter E, Buchler MW, Giese NA, Brors B, Frei C, Murray A, Halama N, Zornig I, Chen YT, Andrews C, Ritter G, Old LJ, Odunsi K, Jager D. Seromic profiling of ovarian and pancreatic cancer. Proc Natl Acad Sci U S A. 2010 Mar 16;107(11):5088-93. doi: 10.1073/pnas.0914213107. Epub 2010 Mar 1. PMID 20194765
- [Background] Mitsuhashi M. Ex vivo simulation of leukocyte function: stimulation of specific subset of leukocytes in whole blood followed by the measurement of function-associated mRNAs. J Immunol Methods. 2010 Dec 15;363(1):95-100. doi: 10.1016/j.jim.2010.10.002. Epub 2010 Oct 15. PMID 20951704
- [Background] Newell EW, Sigal N, Bendall SC, Nolan GP, Davis MM. Cytometry by time-of-flight shows combinatorial cytokine expression and virus-specific cell niches within a continuum of CD8+ T cell phenotypes. Immunity. 2012 Jan 27;36(1):142-52. doi: 10.1016/j.immuni.2012.01.002. PMID 22265676
- [Background] Bogunovic D, O'Neill DW, Belitskaya-Levy I, Vacic V, Yu YL, Adams S, Darvishian F, Berman R, Shapiro R, Pavlick AC, Lonardi S, Zavadil J, Osman I, Bhardwaj N. Immune profile and mitotic index of metastatic melanoma lesions enhance clinical staging in predicting patient survival. Proc Natl Acad Sci U S A. 2009 Dec 1;106(48):20429-34. doi: 10.1073/pnas.0905139106. Epub 2009 Nov 13. PMID 19915147
- [Background] Nair SS…. Salazar A, Galsky M, Bhardwaj N and Tewari A. Phase I study of in situ autologous vaccination for prostate cancer in a neo-adjuvant setting [abstract]. In: Proceedings of the American Association for Cancer Research Annual Meeting 2019; 2019 Mar 29-Apr 3; Atlanta, GA. Philadelphia (PA): AACR; Cancer Res 2019;79(13 Suppl):Abstract nr CT096